CLINICAL TRIAL: NCT01790035
Title: A Phase I and Randomized Controlled Phase II Trial of the Probiotic LGG for Prevention of Side Effects in Patients Undergoing Chemoradiation for Gastrointestinal Cancer
Brief Title: Probiotic LGG for Prevention of Side Effects in Patients Undergoing Chemoradiation for Gastrointestinal Cancer
Acronym: LGG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201404101
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Gastrointestinal Neoplasms
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LGG (Experimental): LGG (containing 10^10 viable bacteria) taken by mouth twice daily beginning at baseline (but starting at least 3 days prior to the start of radiation) and continue during RT and for the 2 weeks following RT.
  Interventions: Drug: LGG
- Placebo (Experimental): Placebo taken by mouth twice daily beginning at baseline (but starting at least 3 days prior to the start of radiation) and continue during RT and for the 2 weeks following RT.
  Interventions: Drug: Placebo
- No intervention (No Intervention): Patients who prefer not to receive LGG will not be randomized and will receive standard of care RT. These patients will serve as a non-intervention comparator cohort to the first 20 patients and will have specimens collected but will not receive the placebo.

INTERVENTIONS:
Drug: LGG
  Other Names: Culturelle
  Arms: LGG
Drug: Placebo
  Arms: Placebo

SUMMARY:
Phase 3 placebo-controlled trial to determine efficacy of the probiotic LGG for reducing acute treatment related GI toxicity in patients with GI malignancy with phase 1 safety lead-in.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of a gastrointestinal, abdominal, or pelvic cancer for which the use of continuous definitive or adjuvant external-beam RT to the abdomen or pelvis to a minimum dose of 4500 cGy is planned.
* Scheduled to receive concurrent administration of fluoropyrimidine chemotherapy (5-FU or capecitabine) during radiation therapy.
* Age ≥ 18 years.
* Life expectancy ≥ 6 months.
* Negative pregnancy test done ≤7 days prior to registration (for women of childbearing potential only).
* The following laboratory values obtained ≤ 28 days prior to registration:

  * Hemoglobin ≥ 9.0 g/dL
  * WBC ≥ 3,500
  * Absolute neutrophil count ≥ 1,500
  * Platelets ≥ 100,000
* ECOG Performance Status (PS) of 0, 1, or 2.
* Willingness to abstain from ingestion of yogurt products and/or any product containing probiotics during study drug treatment.
* Ability to complete questionnaire(s) alone or with assistance.
* Ability to understand and willingness to sign informed consent.

Exclusion Criteria:

* Previous bowel resection which, in the opinion of the investigator, would decrease the benefit of the probiotic. Patients who have undergone recent bowel surgeries which would not decrease the benefit of the probiotic are eligible provided they are more than 30 days from surgery with no serious complications.
* Known allergy to a probiotic preparation.
* Any history of inflammatory bowel disease.
* Grade 3 or 4 diarrhea, rectal bleeding, abdominal cramping, or incontinence of stool ≤7 days prior to registration.
* Any medical condition that may interfere with ability to receive protocol treatment.
* Prior abdominal or pelvic RT.
* Use of probiotics ≤ 2 weeks prior to registration.
* Use of antibiotics ≤ 3 days prior to registration.
* Planned continuous antibiotic treatment during RT.
* History of gastrointestinal or genitourinary obstruction or porphyria.
* History of irritable bowel syndrome (IBS).
* History of hypersensitivity to all of the following antibiotics: penicillin, erythromycin, clindamycin, and any fluoroquinolone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Efficacy (randomized phase II trial) | Up to 6 months following the last dose of LGG or placebo
  Compare the proportion of patients receiving abdominal or pelvic chemoradiation with a fluoropyrimidine being treated with the probiotic LGG who develop CTCAE grade 2 or greater diarrhea to the proportion of patients receiving abdominal or pelvic chemoradiation with a fluoropyrimidine being treated with placebo who develop CTCAE grade 2 or greater diarrhea
Safety (phase I safety lead-in) | Up to 30 days following completion of treatment
  Determine the safety and tolerability of LGG in patients receiving abdominal or pelvic chemoradiation with a fluoropyrimidine
  The DSMC will review the data as part of an interim analysis when the last patient has had 30 days of follow-up. The DSMC will ensure that at least 18 patients have had follow-up at 30 days (with expected 10% drop-out). Accrual to the randomized portion of the trial will occur only if there are no episodes of lactobacillus associated septicemia. Additionally, if two or more serious adverse events of a similar nature occur and a causal relationship to the investigational product cannot be excluded, accrual to the randomized portion will not occur.

SECONDARY OUTCOMES:
Diarrhea subscale score | Up to 5 years after completion of treatment.
  The average AUC of the FACIT-D diarrhea subscale scores will be compared between the two treatment groups using a two-sample t-test.
  The FACIT-D will be completed at baseline, weekly during radiation treatment, for the two weeks following completion of radiation treatment, 12 months following the end of radiation treatment, and years 2-5 following the completion of radiation treatment.
Need for antidiarrhea medication | Up to 2 weeks after completion of treatment
  Need for use of an antidiarrheal medication (Loperamide) will be evaluated at a binary endpoint (Use or No Use). Comparison will be made using Fisher's exact test as previously described (Chitapanarux 2010)
Grade 3 or greater diarrhea | Up to 6 months following the last dose of LGG or placebo
  In patients receiving abdominal or pelvic chemoradiation with a fluoropyrimidine, compare the proportion of patients who develop diarrhea of grade 3 or greater (by CTCAE version 4.0) in those treated with the probiotic LGG to the proportion in those receiving placebo
Fecal calprotectin | Up to 2 weeks following the completion of treatment
  Determine whether fecal calprotectin correlates with onset, duration, and/or severity of diarrhea during chemoradiation
Serum citrulline | Up to 2 weeks following the completion of treatment
  Determine whether serum citrulline correlates with onset, duration, and/or severity of diarrhea during chemoradiation

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ciorba, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Packey CD, Ciorba MA. Microbial influences on the small intestinal response to radiation injury. Curr Opin Gastroenterol. 2010 Mar;26(2):88-94. doi: 10.1097/MOG.0b013e3283361927. PMID 20040865
- [Background] Ciorba MA, Stenson WF. Probiotic therapy in radiation-induced intestinal injury and repair. Ann N Y Acad Sci. 2009 May;1165:190-4. doi: 10.1111/j.1749-6632.2009.04029.x. PMID 19538306
- [Background] Chitapanarux I, Chitapanarux T, Traisathit P, Kudumpee S, Tharavichitkul E, Lorvidhaya V. Randomized controlled trial of live lactobacillus acidophilus plus bifidobacterium bifidum in prophylaxis of diarrhea during radiotherapy in cervical cancer patients. Radiat Oncol. 2010 May 5;5:31. doi: 10.1186/1748-717X-5-31. PMID 20444243
- [Background] Ciorba MA, Riehl TE, Rao MS, Moon C, Ee X, Nava GM, Walker MR, Marinshaw JM, Stappenbeck TS, Stenson WF. Lactobacillus probiotic protects intestinal epithelium from radiation injury in a TLR-2/cyclo-oxygenase-2-dependent manner. Gut. 2012 Jun;61(6):829-38. doi: 10.1136/gutjnl-2011-300367. Epub 2011 Oct 24. PMID 22027478
- [Derived] Riehl TE, Alvarado D, Ee X, Zuckerman A, Foster L, Kapoor V, Thotala D, Ciorba MA, Stenson WF. Lactobacillus rhamnosus GG protects the intestinal epithelium from radiation injury through release of lipoteichoic acid, macrophage activation and the migration of mesenchymal stem cells. Gut. 2019 Jun;68(6):1003-1013. doi: 10.1136/gutjnl-2018-316226. Epub 2018 Jun 22. PMID 29934438
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu